CLINICAL TRIAL: NCT01839461
Title: Personalizing Perioperative Morphine Analgesia for Adolescents Undergoing Major Spine Surgeries
Brief Title: Pharmacogenetic Morphine Spine Study
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0973
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: Pharmacogenetics; postoperative; pediatric; opioid; perioperative; respiratory depression; chronic pain
MeSH Terms: conditions — Pain; Respiratory Insufficiency; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — De-identified study subjects' genetic information and their responses to pain and pain medications, side-effects will be included in a study database. No patient identifiers will be included in the database and there will be a confidential (access limited to investigators only) code or link between the database and other information about the participant. Repeat timed blood samples will be collected using a sparse sampling strategy to evaluate morphine and metabolite concentrations. DNA from preoperative blood samples will be analyzed using genetic and epigenetic arrays, as well plasma for inflammatory markers.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to identify factors and genes (the DNA material that determines the makeup of the human body) that may be associated with how children cope with pain and respond to pain medication. Morphine is a pain medication commonly prescribed after this surgery during the hospital stay. The investigators want to study factors that may be associated with morphine requirement after surgery and side-effects from morphine. They will use pharmacometric models to identify dosing guidelines and factors associated with individual variability in metabolism and efficacy/safety of morphine. They will also study psychological, genetic and epigenetic factors associated with acute and chronic post-surgical pain after spine surgery. The investigators expect that the information obtained in this research study will help to develop effective, safer, and tailored treatment options in the future.

DETAILED DESCRIPTION:
Safe and effective analgesia is an important unmet medical need in children. Despite efforts to promote non-pharmacologic interventions, drug treatment remains the standard of care for children experiencing severe pain following surgery. Inadequate pain relief after invasive surgery, and side effects from analgesics such as morphine occur frequently in up to 50% of children. A study of patient-controlled analgesia morphine use after spine surgery in adolescents observed a 45% incidence of postoperative nausea and vomiting 15% incidence of pruritis and 7% incidence of respiratory depression. Among the drugs available, the opioids, specifically morphine is the most commonly employed. Morphine has a narrow therapeutic index, with the most fatal toxicity being respiratory depression. For morphine, like most opioids, there is a fine balance in dosing regimen between optimal pain control and safety in terms of decreasing morphine's respiratory depressant/ sedative side effects. Inadequate pain relief and analgesic side effects have major clinical, behavioral and economic consequences. Neither evidence-based dosing guidelines nor rigorous documentation of therapeutic benefit for morphine has been ascertained in the pediatric patient population. Despite aggressive pain management after spine surgery, findings showed that neither children's pain nor their analgesic use diminished significantly over time. As such, there is a critical knowledge gap in the medical literature that significantly impacts the pediatric pain management. In recognition of this therapeutic challenge the investigators plan to evaluate the determinants of inter-individual differences in opioid analgesic responsiveness and adverse effects in children. Adolescents following spine surgery have a great variability in morphine requirements with greater use as they became older. Analgesic dosing is dependent on appreciation of the interplay between pharmacokinetics, pharmacodynamics and therapeutics. These factors are often poorly understood, where the effective control of procedural pain for example, remains problematic. Suitable pharmacological alternatives to opioid treatment for moderate to severe pain in children after surgery are limited and consequently there is a need for a critical evaluation of the existing opioids and research reports.

Recently a number of small studies have shown the association of single nucleotide polymorphism in genes in the pain pathway, with altered pain response to a stimulus or altered response to opioids following a painful procedure. Age, gender, cultural influences, anxiety, type of surgical procedure and genetic factors can all influence the response. By extending follow up of patients to years after surgery, the aims were amended to include evaluation of chronic post-surgical outcomes.

We will be collecting data on pain scores, opioid effects, psychological questionnaires, blood samples and pupillometry data.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10 to 18, inclusive, years of age
* Diagnosis of Idiopathic scoliosis, kyphosis and/or kyphoscoliosis
* Scheduled for spine fusion

Exclusion Criteria:

* Known hypersensitivity to morphine
* Patients on chronic pain medication.
* Pregnant or breastfeeding females.
* Children with a history of or active renal or liver disease.
* Concomitant use of medication known to induce or inhibit CYP2D6 activity including paroxetine, fluoxetine, cimetidine, duloxetine or methadone.
* Non-English speaking patients.
* Developmental delay.
* Children who have problems with pupil or pupillary reaction due to disease (such as amyloidosis, bilateral Horner's syndrome, familial dysautonomia, other major neurological disorders) or preoperative medications influencing pupillary size (anti-cholinergic, narcotic medications such as codeine in cough syrup) will be recruited but pupillometry will be deferred.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children ages 10 to 18, inclusive, years scheduled for spinal surgical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2009-07; Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Immediate postoperative pain scores in the recovery room | 1 day ( Recovery room)
  Pain score will be measured using standard and validated scales, Numeric rating scale (NRS 0 - 10). This scale has been widely validated and discriminates mild, moderate and severe pain

SECONDARY OUTCOMES:
postoperative intravenous morphine requirement | First 48 hours after surgery
  Pain score will be measured using standard and validated scales, Numeric rating scale (NRS 0 - 10). This scale has been widely validated and discriminates mild, moderate and severe pain.
Chronic pain pre-operatively | Pre-operative
  Participants will complete questionnaires regarding pain since surgery was completed
Chronic pain post-operatively | 2 - 6 months post-operative
  Participants will complete questionnaires regarding pain since surgery was completed
Chronic pain post-operatively | 10 - 12 months post-operative
  Participants will complete questionnaires regarding pain since surgery was completed

OTHER OUTCOMES:
Side-effect measures | First 48 hours post surgery
  Incidences of respiratory depression, sedation, postoperative nausea and vomiting (PONV) in the recovery phase will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Chidambaran, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Beaulieu P, Cyrenne L, Mathews S, Villeneuve E, Vischoff D. Patient-controlled analgesia after spinal fusion for idiopathic scoliosis. Int Orthop. 1996;20(5):295-9. doi: 10.1007/s002640050081. PMID 8930721
- [Background] Rahim-Williams FB, Riley JL 3rd, Herrera D, Campbell CM, Hastie BA, Fillingim RB. Ethnic identity predicts experimental pain sensitivity in African Americans and Hispanics. Pain. 2007 May;129(1-2):177-84. doi: 10.1016/j.pain.2006.12.016. Epub 2007 Feb 12. PMID 17296267
- [Background] Rakvag TT, Klepstad P, Baar C, Kvam TM, Dale O, Kaasa S, Krokan HE, Skorpen F. The Val158Met polymorphism of the human catechol-O-methyltransferase (COMT) gene may influence morphine requirements in cancer pain patients. Pain. 2005 Jul;116(1-2):73-8. doi: 10.1016/j.pain.2005.03.032. PMID 15927391
- [Background] Nackley AG, Tan KS, Fecho K, Flood P, Diatchenko L, Maixner W. Catechol-O-methyltransferase inhibition increases pain sensitivity through activation of both beta2- and beta3-adrenergic receptors. Pain. 2007 Apr;128(3):199-208. doi: 10.1016/j.pain.2006.09.022. Epub 2006 Nov 7. PMID 17084978
- [Background] Diatchenko L, Nackley AG, Slade GD, Bhalang K, Belfer I, Max MB, Goldman D, Maixner W. Catechol-O-methyltransferase gene polymorphisms are associated with multiple pain-evoking stimuli. Pain. 2006 Dec 5;125(3):216-224. doi: 10.1016/j.pain.2006.05.024. Epub 2006 Jul 11. PMID 16837133
- [Background] Diatchenko L, Slade GD, Nackley AG, Bhalang K, Sigurdsson A, Belfer I, Goldman D, Xu K, Shabalina SA, Shagin D, Max MB, Makarov SS, Maixner W. Genetic basis for individual variations in pain perception and the development of a chronic pain condition. Hum Mol Genet. 2005 Jan 1;14(1):135-43. doi: 10.1093/hmg/ddi013. Epub 2004 Nov 10. PMID 15537663
- [Background] Zubieta JK, Heitzeg MM, Smith YR, Bueller JA, Xu K, Xu Y, Koeppe RA, Stohler CS, Goldman D. COMT val158met genotype affects mu-opioid neurotransmitter responses to a pain stressor. Science. 2003 Feb 21;299(5610):1240-3. doi: 10.1126/science.1078546. PMID 12595695
- [Background] Oertel BG, Schmidt R, Schneider A, Geisslinger G, Lotsch J. The mu-opioid receptor gene polymorphism 118A>G depletes alfentanil-induced analgesia and protects against respiratory depression in homozygous carriers. Pharmacogenet Genomics. 2006 Sep;16(9):625-36. doi: 10.1097/01.fpc.0000220566.90466.a2. PMID 16906017
- [Background] Chou WY, Wang CH, Liu PH, Liu CC, Tseng CC, Jawan B. Human opioid receptor A118G polymorphism affects intravenous patient-controlled analgesia morphine consumption after total abdominal hysterectomy. Anesthesiology. 2006 Aug;105(2):334-7. doi: 10.1097/00000542-200608000-00016. PMID 16871067
- [Background] Chou WY, Yang LC, Lu HF, Ko JY, Wang CH, Lin SH, Lee TH, Concejero A, Hsu CJ. Association of mu-opioid receptor gene polymorphism (A118G) with variations in morphine consumption for analgesia after total knee arthroplasty. Acta Anaesthesiol Scand. 2006 Aug;50(7):787-92. doi: 10.1111/j.1399-6576.2006.01058.x. PMID 16879459
- [Background] Klepstad P, Rakvag TT, Kaasa S, Holthe M, Dale O, Borchgrevink PC, Baar C, Vikan T, Krokan HE, Skorpen F. The 118 A > G polymorphism in the human mu-opioid receptor gene may increase morphine requirements in patients with pain caused by malignant disease. Acta Anaesthesiol Scand. 2004 Nov;48(10):1232-9. doi: 10.1111/j.1399-6576.2004.00517.x. PMID 15504181
- [Background] Reyes-Gibby CC, Shete S, Rakvag T, Bhat SV, Skorpen F, Bruera E, Kaasa S, Klepstad P. Exploring joint effects of genes and the clinical efficacy of morphine for cancer pain: OPRM1 and COMT gene. Pain. 2007 Jul;130(1-2):25-30. doi: 10.1016/j.pain.2006.10.023. Epub 2006 Dec 6. PMID 17156920
- [Background] Pasternak GW. The pharmacology of mu analgesics: from patients to genes. Neuroscientist. 2001 Jun;7(3):220-31. doi: 10.1177/107385840100700307. PMID 11499401
- [Background] Coulbault L, Beaussier M, Verstuyft C, Weickmans H, Dubert L, Tregouet D, Descot C, Parc Y, Lienhart A, Jaillon P, Becquemont L. Environmental and genetic factors associated with morphine response in the postoperative period. Clin Pharmacol Ther. 2006 Apr;79(4):316-24. doi: 10.1016/j.clpt.2006.01.007. PMID 16580900
- [Background] Coller JK, Barratt DT, Dahlen K, Loennechen MH, Somogyi AA. ABCB1 genetic variability and methadone dosage requirements in opioid-dependent individuals. Clin Pharmacol Ther. 2006 Dec;80(6):682-90. doi: 10.1016/j.clpt.2006.09.011. PMID 17178268
- [Background] Rakvag TT, Ross JR, Sato H, Skorpen F, Kaasa S, Klepstad P. Genetic variation in the catechol-O-methyltransferase (COMT) gene and morphine requirements in cancer patients with pain. Mol Pain. 2008 Dec 18;4:64. doi: 10.1186/1744-8069-4-64. PMID 19094200
- [Background] Gramke HF, de Rijke JM, van Kleef M, Raps F, Kessels AG, Peters ML, Sommer M, Marcus MA. The prevalence of postoperative pain in a cross-sectional group of patients after day-case surgery in a university hospital. Clin J Pain. 2007 Jul-Aug;23(6):543-8. doi: 10.1097/AJP.0b013e318074c970. PMID 17575496
- [Background] Ikeda K, Ide S, Han W, Hayashida M, Uhl GR, Sora I. How individual sensitivity to opiates can be predicted by gene analyses. Trends Pharmacol Sci. 2005 Jun;26(6):311-7. doi: 10.1016/j.tips.2005.04.001. PMID 15925706
- [Background] Ameyaw MM, Regateiro F, Li T, Liu X, Tariq M, Mobarek A, Thornton N, Folayan GO, Githang'a J, Indalo A, Ofori-Adjei D, Price-Evans DA, McLeod HL. MDR1 pharmacogenetics: frequency of the C3435T mutation in exon 26 is significantly influenced by ethnicity. Pharmacogenetics. 2001 Apr;11(3):217-21. doi: 10.1097/00008571-200104000-00005. PMID 11337937
- [Background] Kim RB, Leake BF, Choo EF, Dresser GK, Kubba SV, Schwarz UI, Taylor A, Xie HG, McKinsey J, Zhou S, Lan LB, Schuetz JD, Schuetz EG, Wilkinson GR. Identification of functionally variant MDR1 alleles among European Americans and African Americans. Clin Pharmacol Ther. 2001 Aug;70(2):189-99. doi: 10.1067/mcp.2001.117412. PMID 11503014
- [Background] Kim H, Neubert JK, San Miguel A, Xu K, Krishnaraju RK, Iadarola MJ, Goldman D, Dionne RA. Genetic influence on variability in human acute experimental pain sensitivity associated with gender, ethnicity and psychological temperament. Pain. 2004 Jun;109(3):488-496. doi: 10.1016/j.pain.2004.02.027. PMID 15157710
- [Background] Khasar SG, McCarter G, Levine JD. Epinephrine produces a beta-adrenergic receptor-mediated mechanical hyperalgesia and in vitro sensitization of rat nociceptors. J Neurophysiol. 1999 Mar;81(3):1104-12. doi: 10.1152/jn.1999.81.3.1104. PMID 10085337
- [Background] Diatchenko L, Anderson AD, Slade GD, Fillingim RB, Shabalina SA, Higgins TJ, Sama S, Belfer I, Goldman D, Max MB, Weir BS, Maixner W. Three major haplotypes of the beta2 adrenergic receptor define psychological profile, blood pressure, and the risk for development of a common musculoskeletal pain disorder. Am J Med Genet B Neuropsychiatr Genet. 2006 Jul 5;141B(5):449-62. doi: 10.1002/ajmg.b.30324. PMID 16741943
- [Background] Liang DY, Liao G, Wang J, Usuka J, Guo Y, Peltz G, Clark JD. A genetic analysis of opioid-induced hyperalgesia in mice. Anesthesiology. 2006 May;104(5):1054-62. doi: 10.1097/00000542-200605000-00023. PMID 16645459
- [Background] Coffman BL, Rios GR, King CD, Tephly TR. Human UGT2B7 catalyzes morphine glucuronidation. Drug Metab Dispos. 1997 Jan;25(1):1-4. PMID 9010622
- [Background] Hirota T, Ieiri I, Takane H, Sano H, Kawamoto K, Aono H, Yamasaki A, Takeuchi H, Masada M, Shimizu E, Higuchi S, Otsubo K. Sequence variability and candidate gene analysis in two cancer patients with complex clinical outcomes during morphine therapy. Drug Metab Dispos. 2003 May;31(5):677-80. doi: 10.1124/dmd.31.5.677. PMID 12695358
- [Background] Duguay Y, Baar C, Skorpen F, Guillemette C. A novel functional polymorphism in the uridine diphosphate-glucuronosyltransferase 2B7 promoter with significant impact on promoter activity. Clin Pharmacol Ther. 2004 Mar;75(3):223-33. doi: 10.1016/j.clpt.2003.10.006. PMID 15001974
- [Background] Takeda S, Ishii Y, Iwanaga M, Mackenzie PI, Nagata K, Yamazoe Y, Oguri K, Yamada H. Modulation of UDP-glucuronosyltransferase function by cytochrome P450: evidence for the alteration of UGT2B7-catalyzed glucuronidation of morphine by CYP3A4. Mol Pharmacol. 2005 Mar;67(3):665-72. doi: 10.1124/mol.104.007641. Epub 2004 Dec 20. PMID 15611481
- [Background] Smith HS. Opioid metabolism. Mayo Clin Proc. 2009 Jul;84(7):613-24. doi: 10.1016/S0025-6196(11)60750-7. PMID 19567715
- [Background] Schaffer JV, Bolognia JL. The melanocortin-1 receptor: red hair and beyond. Arch Dermatol. 2001 Nov;137(11):1477-85. doi: 10.1001/archderm.137.11.1477. PMID 11708951
- [Background] Mogil JS, Wilson SG, Chesler EJ, Rankin AL, Nemmani KV, Lariviere WR, Groce MK, Wallace MR, Kaplan L, Staud R, Ness TJ, Glover TL, Stankova M, Mayorov A, Hruby VJ, Grisel JE, Fillingim RB. The melanocortin-1 receptor gene mediates female-specific mechanisms of analgesia in mice and humans. Proc Natl Acad Sci U S A. 2003 Apr 15;100(8):4867-72. doi: 10.1073/pnas.0730053100. Epub 2003 Mar 27. PMID 12663858
- [Background] Mogil JS, Ritchie J, Smith SB, Strasburg K, Kaplan L, Wallace MR, Romberg RR, Bijl H, Sarton EY, Fillingim RB, Dahan A. Melanocortin-1 receptor gene variants affect pain and mu-opioid analgesia in mice and humans. J Med Genet. 2005 Jul;42(7):583-7. doi: 10.1136/jmg.2004.027698. PMID 15994880
- [Background] Beaumont KA, Newton RA, Smit DJ, Leonard JH, Stow JL, Sturm RA. Altered cell surface expression of human MC1R variant receptor alleles associated with red hair and skin cancer risk. Hum Mol Genet. 2005 Aug 1;14(15):2145-54. doi: 10.1093/hmg/ddi219. Epub 2005 Jun 22. PMID 15972726
- [Background] Crawford MW, Hickey C, Zaarour C, Howard A, Naser B. Development of acute opioid tolerance during infusion of remifentanil for pediatric scoliosis surgery. Anesth Analg. 2006 Jun;102(6):1662-7. doi: 10.1213/01.ane.0000216036.95705.c2. PMID 16717305
- [Background] Angst MS, Koppert W, Pahl I, Clark DJ, Schmelz M. Short-term infusion of the mu-opioid agonist remifentanil in humans causes hyperalgesia during withdrawal. Pain. 2003 Nov;106(1-2):49-57. doi: 10.1016/s0304-3959(03)00276-8. PMID 14581110
- [Background] Vinik HR, Kissin I. Rapid development of tolerance to analgesia during remifentanil infusion in humans. Anesth Analg. 1998 Jun;86(6):1307-11. doi: 10.1097/00000539-199806000-00033. PMID 9620525
- [Background] Li X, Angst MS, Clark JD. A murine model of opioid-induced hyperalgesia. Brain Res Mol Brain Res. 2001 Jan 31;86(1-2):56-62. doi: 10.1016/s0169-328x(00)00260-6. PMID 11165371
- [Background] Mao J, Sung B, Ji RR, Lim G. Chronic morphine induces downregulation of spinal glutamate transporters: implications in morphine tolerance and abnormal pain sensitivity. J Neurosci. 2002 Sep 15;22(18):8312-23. doi: 10.1523/JNEUROSCI.22-18-08312.2002. PMID 12223586
- [Background] King T, Gardell LR, Wang R, Vardanyan A, Ossipov MH, Malan PT Jr, Vanderah TW, Hunt SP, Hruby VJ, Lai J, Porreca F. Role of NK-1 neurotransmission in opioid-induced hyperalgesia. Pain. 2005 Aug;116(3):276-288. doi: 10.1016/j.pain.2005.04.014. PMID 15964684
- [Background] Moises HC, Smith CB. Changes occur in central adrenoreceptor function following long-term morphine treatment and during morphine withdrawal. Neuropeptides. 1984 Dec;5(1-3):29-32. doi: 10.1016/0143-4179(84)90019-2. PMID 6152326
- [Background] Hood DD, Curry R, Eisenach JC. Intravenous remifentanil produces withdrawal hyperalgesia in volunteers with capsaicin-induced hyperalgesia. Anesth Analg. 2003 Sep;97(3):810-815. doi: 10.1213/01.ANE.0000078811.80093.88. PMID 12933407
- [Background] Nackley A, Diatchenko L, Maixner W. Perspectives on the genetic basis of opioid-induced hyperalgesia. Anesthesiology. 2006 May;104(5):909-10. doi: 10.1097/00000542-200605000-00004. No abstract available. PMID 16645440
- [Background] Perquin CW, Hazebroek-Kampschreur AAJM, Hunfeld JAM, Bohnen AM, van Suijlekom-Smit LWA, Passchier J, van der Wouden JC. Pain in children and adolescents: a common experience. Pain. 2000 Jul;87(1):51-58. doi: 10.1016/S0304-3959(00)00269-4. PMID 10863045
- [Background] Duedahl TH, Hansen EH. A qualitative systematic review of morphine treatment in children with postoperative pain. Paediatr Anaesth. 2007 Aug;17(8):756-74. doi: 10.1111/j.1460-9592.2007.02213.x. PMID 17596221
- [Background] Anderson BJ, Palmer GM. Recent developments in the pharmacological management of pain in children. Curr Opin Anaesthesiol. 2006 Jun;19(3):285-92. doi: 10.1097/01.aco.0000192802.33291.6f. PMID 16735812
- [Background] Klepstad P, Dale O, Skorpen F, Borchgrevink PC, Kaasa S. Genetic variability and clinical efficacy of morphine. Acta Anaesthesiol Scand. 2005 Aug;49(7):902-8. doi: 10.1111/j.1399-6576.2005.00772.x. PMID 16045647
- [Background] Berde CB, Sethna NF. Analgesics for the treatment of pain in children. N Engl J Med. 2002 Oct 3;347(14):1094-103. doi: 10.1056/NEJMra012626. No abstract available. PMID 12362012
- [Background] Kotzer AM, Foster R. Children's use of PCA following spinal fusion. Orthop Nurs. 2000 Sep-Oct;19(5):19-27; quiz 28-30. doi: 10.1097/00006416-200019050-00005. PMID 11153382
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Gibson PR. Anaesthesia for correction of scoliosis in children. Anaesth Intensive Care. 2004 Aug;32(4):548-59. doi: 10.1177/0310057X0403200413. PMID 15675216
- [Background] Hong D, Flood P, Diaz G. The side effects of morphine and hydromorphone patient-controlled analgesia. Anesth Analg. 2008 Oct;107(4):1384-9. doi: 10.1213/ane.0b013e3181823efb. PMID 18806056
- [Background] Sadhasivam S, Cohen LL, Szabova A, Varughese A, Kurth CD, Willging P, Wang Y, Nick TG, Gunter J. Real-time assessment of perioperative behaviors and prediction of perioperative outcomes. Anesth Analg. 2009 Mar;108(3):822-6. doi: 10.1213/ane.0b013e318195c115. PMID 19224789
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Chen E, Zeltzer LK, Craske MG, Katz ER. Alteration of memory in the reduction of children's distress during repeated aversive medical procedures. J Consult Clin Psychol. 1999 Aug;67(4):481-90. doi: 10.1037//0022-006x.67.4.481. PMID 10450618
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] von Baeyer CL. Numerical rating scale for self-report of pain intensity in children and adolescents: recent progress and further questions. Eur J Pain. 2009 Nov;13(10):1005-7. doi: 10.1016/j.ejpain.2009.08.006. Epub 2009 Sep 17. No abstract available. PMID 19766028
- [Background] von Baeyer CL, Spagrud LJ, McCormick JC, Choo E, Neville K, Connelly MA. Three new datasets supporting use of the Numerical Rating Scale (NRS-11) for children's self-reports of pain intensity. Pain. 2009 Jun;143(3):223-227. doi: 10.1016/j.pain.2009.03.002. Epub 2009 Apr 8. PMID 19359097
- [Background] Bulloch B, Tenenbein M. Validation of 2 pain scales for use in the pediatric emergency department. Pediatrics. 2002 Sep;110(3):e33. doi: 10.1542/peds.110.3.e33. PMID 12205283
- [Background] Voepel-Lewis T, Marinkovic A, Kostrzewa A, Tait AR, Malviya S. The prevalence of and risk factors for adverse events in children receiving patient-controlled analgesia by proxy or patient-controlled analgesia after surgery. Anesth Analg. 2008 Jul;107(1):70-5. doi: 10.1213/ane.0b013e318172fa9e. PMID 18635469
- [Background] Kharasch ED, Hoffer C, Whittington D, Sheffels P. Role of hepatic and intestinal cytochrome P450 3A and 2B6 in the metabolism, disposition, and miotic effects of methadone. Clin Pharmacol Ther. 2004 Sep;76(3):250-69. doi: 10.1016/j.clpt.2004.05.003. PMID 15371986
- [Background] Kharasch ED, Walker A, Hoffer C, Sheffels P. Intravenous and oral alfentanil as in vivo probes for hepatic and first-pass cytochrome P450 3A activity: noninvasive assessment by use of pupillary miosis. Clin Pharmacol Ther. 2004 Nov;76(5):452-66. doi: 10.1016/j.clpt.2004.07.006. PMID 15536460
- [Background] Constant I, Nghe MC, Boudet L, Berniere J, Schrayer S, Seeman R, Murat I. Reflex pupillary dilatation in response to skin incision and alfentanil in children anaesthetized with sevoflurane: a more sensitive measure of noxious stimulation than the commonly used variables. Br J Anaesth. 2006 May;96(5):614-9. doi: 10.1093/bja/ael073. Epub 2006 Mar 24. PMID 16565227
- [Background] Boev AN, Fountas KN, Karampelas I, Boev C, Machinis TG, Feltes C, Okosun I, Dimopoulos V, Troup C. Quantitative pupillometry: normative data in healthy pediatric volunteers. J Neurosurg. 2005 Dec;103(6 Suppl):496-500. doi: 10.3171/ped.2005.103.6.0496. PMID 16383247
- [Background] Gozal D, Ben-Ari JH, Harper RM, Keens TG. Ventilatory responses to repeated short hypercapnic challenges. J Appl Physiol (1985). 1995 Apr;78(4):1374-81. doi: 10.1152/jappl.1995.78.4.1374. PMID 7615445
- [Background] Ross JR, Rutter D, Welsh K, Joel SP, Goller K, Wells AU, Du Bois R, Riley J. Clinical response to morphine in cancer patients and genetic variation in candidate genes. Pharmacogenomics J. 2005;5(5):324-36. doi: 10.1038/sj.tpj.6500327. PMID 16103897
- [Background] Cepeda MS, Farrar JT, Baumgarten M, Boston R, Carr DB, Strom BL. Side effects of opioids during short-term administration: effect of age, gender, and race. Clin Pharmacol Ther. 2003 Aug;74(2):102-12. doi: 10.1016/S0009-9236(03)00152-8. PMID 12891220
- [Background] Kelly PJ, Stallard N, Whittaker JC. Statistical design and analysis of pharmacogenetic trials. Stat Med. 2005 May 30;24(10):1495-508. doi: 10.1002/sim.2052. PMID 15706636
- [Background] Musani SK, Shriner D, Liu N, Feng R, Coffey CS, Yi N, Tiwari HK, Allison DB. Detection of gene x gene interactions in genome-wide association studies of human population data. Hum Hered. 2007;63(2):67-84. doi: 10.1159/000099179. Epub 2007 Feb 2. PMID 17283436
- [Background] Gardiner JC, Luo Z, Roman LA. Fixed effects, random effects and GEE: what are the differences? Stat Med. 2009 Jan 30;28(2):221-39. doi: 10.1002/sim.3478. PMID 19012297
- [Derived] Einhorn LM, Monitto CL, Ganesh A, Duan Q, Lee J, Ramamurthi RJ, Barnett K, Ding L, Chidambaran V. Multi-Institutional Study of Multimodal Analgesia Practice, Pain Trajectories, and Recovery Trends After Spine Fusion for Idiopathic Scoliosis. Anesth Analg. 2025 Nov 1;141(5):1137-1148. doi: 10.1213/ANE.0000000000007351. Epub 2025 Jan 2. PMID 39745877
- [Derived] Chidambaran V, Zhang X, Pilipenko V, Chen X, Wronowski B, Geisler K, Martin LJ, Barski A, Weirauch MT, Ji H. Methylation quantitative trait locus analysis of chronic postsurgical pain uncovers epigenetic mediators of genetic risk. Epigenomics. 2021 Apr;13(8):613-630. doi: 10.2217/epi-2020-0424. Epub 2021 Apr 6. PMID 33820434
- [Derived] Chidambaran V, Ding L, Moore DL, Spruance K, Cudilo EM, Pilipenko V, Hossain M, Sturm P, Kashikar-Zuck S, Martin LJ, Sadhasivam S. Predicting the pain continuum after adolescent idiopathic scoliosis surgery: A prospective cohort study. Eur J Pain. 2017 Aug;21(7):1252-1265. doi: 10.1002/ejp.1025. Epub 2017 Mar 27. PMID 28346762
- [Derived] Chidambaran V, Venkatasubramanian R, Zhang X, Martin LJ, Niu J, Mizuno T, Fukuda T, Meller J, Vinks AA, Sadhasivam S. ABCC3 genetic variants are associated with postoperative morphine-induced respiratory depression and morphine pharmacokinetics in children. Pharmacogenomics J. 2017 Mar;17(2):162-169. doi: 10.1038/tpj.2015.98. Epub 2016 Jan 26. PMID 26810133